CLINICAL TRIAL: NCT00340639
Title: Developmental Influences on Management of Type I Diabetes
Brief Title: Management of Type 1 Diabetes Among Adolescents
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903088; 03-CH-N088
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-11-02

CONDITIONS: Type I Diabetes
Keywords: Adherence; Chronic Illness; Adolescent; Family; Self-Regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Chronic Disease; Self-Control

SUMMARY:
This 1-year study will explore the influences of family and peers on how diabetic adolescents manage their disease, focusing on adolescent developmental transitions. The management of diabetes is a complex process involving daily self-care activities, problem-solving, and decision-making. It is particularly challenging during adolescence when youth are experiencing physiological, social and psychological changes, and coming under increasing peer influence and decreasing parental supervision. Although it is expected that the responsibility for diabetes management will gradually shift from the parent to the child during adolescence, research indicates that many children may be given responsibility for managing their illness too early, without adequate parental monitoring. Specifically, this study will examine the following issues:

* The relationship of peers, parents and school support to successful diabetes management;
* The influence of the adolescent's self-image and personal goals on diabetes management;
* The influence of the adolescent's and parents' attitudes, capability and environment on the balance of responsibility for diabetes management.

Children between 10 and 16 years of age receiving treatment for diabetes type 1 at Georgetown University Medical Center's pediatric diabetes clinic may be eligible for this study. The children must have been diagnosed with diabetes at least 1 year before entering the study and must require insulin treatment. One parent of each child will also participate in the study.

Children and their parents will complete the following procedures:

Home Interviews: Parents and children will complete two at-home face-to-face interviews 6 months apart. At each interview, children will answer questions about their responsibility for and adherence to their diabetes management, treatment outcome expectations, optimism, self-esteem, self-consciousness, personal goals, social support, perceived barriers to diabetes management, family routine and family conflict, their parents' involvement in their diabetes management, and parenting style. Parents will evaluate their child's ability to manage his or her diabetes, level of maturity, self-esteem, and transition of responsibility; their family routine and family conflict, parent-child communication, their parenting goals, and their involvement in and responsibility for their child's diabetes management. Three days after the 6-month interview, a randomly selected group of parents and children will complete a brief, additional telephone interview covering some of the same issues.

Telephone Interview: At 12 months, parents and children will complete a telephone interview that will include questions about adherence to diabetes management and the responsibility of parents and children for diabetes management.

DETAILED DESCRIPTION:
Management of diabetes is a complex process involving the conduct of daily self-care activities, problem-solving, and decision-making. It is particularly challenging during adolescence when youth are experiencing a variety of physiological, social, and psychological changes at the same time that they are taking increased responsibility for their own diabetes care. This study examines the influence of family, social, and adolescent developmental transitions. Over the course of 12 months, a sample of 135 parent-child dyads will provide information on individual efficacy, maturity, family and social support, attitudes toward diabetes management, and diabetes management behaviors. One goal of this pilot study is to identify factors that predict the adherence of individual youth and parents during this transition period.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Subjects for this study will include 135 male and female youth with diabetes age 10-16 and a parent.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2003-01-28; Study Completion 2006-11-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson B, Ho J, Brackett J, Finkelstein D, Laffel L. Parental involvement in diabetes management tasks: relationships to blood glucose monitoring adherence and metabolic control in young adolescents with insulin-dependent diabetes mellitus. J Pediatr. 1997 Feb;130(2):257-65. doi: 10.1016/s0022-3476(97)70352-4. PMID 9042129